CLINICAL TRIAL: NCT06801249
Title: "Effect of Metyrapone on Cardiovascular Risk Factors in Patients With Adrenal Incidentalomas and Subclinical/Mild Cushing's Syndrome
Brief Title: Effect of Metyrapone on Cardiovascular Risk Factors in Patients With Adrenal Incidentalomas and Cushing's Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR-MET-19
Record Dates: First submitted 2024-12-01; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Adrenal Incidentalomas; Cushing Syndrome
MeSH Terms: conditions — Adrenal incidentaloma; Cushing Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Metirapone in addition to standardized antihypertensive therapy, as provided in the normal course of care and in accordance with current European guidelines. Metirapone will be provided in 250-mg capsules, in the form of commercially available packs. In Group A, patients will receive Metirapone at the initial dosage of 250 mg, 1 capsule per day. Dosage may be adjusted according to clinical response and tolerability, up to a maximum of 750 mg (3 capsules per day). The drug should be taken after a meal. The drug should be stored at room temperature. The expected duration of study treatment is 12 months, after which patients will discontinue Metirapone and continue with therapies as per the normal course of care.
  Interventions: Drug: Metarapone
- Group B (Active Comparator): Standardized antihypertensive therapy, as provided in the normal course of care and in accordance with current European guidelines.
  Interventions: Drug: Standardized antihypertensive therapy

INTERVENTIONS:
Drug: Metarapone — Metirapone is an inhibitor of the enzyme 11-β-adrenal hydroxylase, which is deputed to catalyze the conversion of 11-desoxycortisol (11-S) to cortisol and 11-deoxycorticosterone (DOC) to corticosterone.
  Arms: Group A
Drug: Standardized antihypertensive therapy — Standardized antihypertensive therapy, as provided in the normal course of care and in accordance with current European guidelines.
  Arms: Group B

SUMMARY:
Drug interventional, controlled, randomized open-label, parallel-group, multicenter study in patients with bilateral adrenal incidentalomas associated with subclinical Cushing's syndrome

DETAILED DESCRIPTION:
Drug interventional, controlled, randomized open-label, parallel-group, multicenter (3 centers in total), interventional study in patients with bilateral adrenal incidentalomas associated with SCS.

The study has 3 phases: run-in (phase 1), randomization (phase 2), and interventional phase (phase 3).

Phase 1. During run-in, patients will receive standardized antihypertensive therapy, as provided in the normal course of care and in accordance with current European guidelines. Four classes of antihypertensives will be used: Angiotensin-Converting Enzyme inhibitors (ACEi) or angiotesnine receptor antagonists (ARBs), calcium channel blockers, thiazide diuretics, and beta-blockers with vasodilator properties (Carvedilol or Nebivolol). Treatment will be chosen according to the recommendations of European guidelines and the patient's clinical condition. Patients will be evaluated monthly to check BP and to identify the lowest effective dose of antihypertensive to maintain BP <130/85 mmHg. BP will be measured during medical visits. Home PA monitoring will also be performed during the 7 days before each medical visit. Echocardiogram, electrocardiogram, 24-hour Holter PA, carotid echodoppler, albumin/creatinine ratio, and indices of glucose and lipid metabolism will also be performed, according to the normal procedures of routine clinical practice performed in patients with this problem. The run-in period will be prolonged until pressor values are stabilized (BP >100/60 mmHg and <130/85 mmHg, under minimal effective dose of antihypertensive therapy), with a minimum duration of 2 months and a maximum of 6 months. If stabilization of blood pressure values (according to the criteria outlined above) is not obtained by the sixth month after enrollment, the run-in period may be extended to a maximum of 10 months. If stabilization of the pressor values (according to the criteria outlined above) is not obtained by that time, the patient will be excluded from the study.

Phase 2. After run-in, patients will be randomized (1:1) to treatment with Metirapone (Group A) or observation (Group B) by computer-generated random sequence.

Phase 3. During the interventional phase, patients (Group A and Group B) will be seen every 4 weeks (+/- 7 days). In addition, patients receiving Metirapone (Group A) will be evaluated every 7 days (+/- 2 days) during the first month to titrate Metirapone according to cortisol and cortisone values, monitor electrolytes, and analyze potential side effects. In some patients, titration of Metirapone up to the maximum tolerated dose (and in any case no more than 750 mg/day) may be prolonged beyond 4 weeks. In this case, weekly visits will continue until the maximum tolerated dose is reached (and in any case no more than 750 mg/day) for a period of up to 4 months, after which the achieved dose of Metirapone will be maintained. Patients assigned to Metirapone treatment will not be allowed to take Paracetamol, Phenytoin and estrogen during the interventional phase. Ambulatory and home PA will be assessed monthly to optimize antihypertensive treatment to maintain PA values <130/85 mmHg. Hypotension (BP <100/60 mmHg) will be treated with modification of antihypertensive therapy. At the end of the interventional phase, cardiovascular and metabolic reevaluation will be performed.

Blood samples for serum and plasma collection will be collected after fasting from the previous evening, before randomization and at the end of the study. Saliva samples will be collected during the entire day before blood collection at 10 predetermined times. Blood samples will be collected monthly in patients treated with Metirapone. Serum and saliva will be used for steroid profiles by LC-MS/MS. The following steroids will be measured: cortisol, 21-desoxycortisol, 11-DF, 17-hydroxyprogesterone (17OHP), Delta4-androstenedione, DHEA, testosterone, progesterone, cortisone, DOC and corticosterone. Cortisol, cortisone, 17OHP, Delta4-androstenedione, DHEA and testosterone will be measured in saliva. Waist circumference and body mass index will be assessed at each visit.

Within 6 months after completion of the study, an abdominal CT scan will be repeated. This investigation will be performed as part of the patients' normal course of care, which involves performing follow-up abdomen CT scans periodically (every 18-36 months).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria - run-in (phase 1)

* Unilateral or bilateral adrenal nodules with benign features associated with thickening of the adrenal arms >5 mm on abdominal CT scan
* SCS (detected 2 times in the 6 months before run-in) defined by the absence of catabolic signs of Cushing's syndrome in association with any of these 3 conditions:

  * Cortisol levels after dexamethasone 1 mg test >50 nmol/L associated with baseline ACTH <10 pg/mL
  * Cortisol levels after dexamethasone 1 mg test >50 nmol/L associated with increased nocturnal (11 pm) salivary cortisol
  * Cortisol levels after dexamethasone 1 mg test >138 nmol/L
* Hypertension (BP ≥140/90 mmHg and/or ongoing antihypertensive treatment)
* Patients who cannot undergo surgery
* Acquisition of informed consent.

Inclusion criteria - randomization (phase 2)

- BP >100/60 mmHg and <130/85 mmHg on antihypertensive therapy (lowest effective dose) within 6-10 months after enrollment.

Exclusion Criteria:

* Body mass index ≥40 kg/m2
* Pregnant or lactating women; diagnosis of pregnancy will be made by serum β-HCG assay
* Women of childbearing age using contraceptive measures other than barrier contraception. Barrier contraceptive measures are: o Male or female condom with or without spermicide o Cervical cup, diaphragm or sponges with spermicide o Combination of male condom and cervical cup, diaphragm or sponges with spermicide (dual barrier methods)
* Treatment with steroids in the last year before enrollment
* Taking medications known to interfere with Metirapone
* Known or suspected hypersensitivity to the drug or drug class under study
* Patients with serious clinical conditions that, in the opinion of the Investigator, contraindicate the patient's participation in the study
* Patients with primary corticosurrenal insufficiency, impaired adrenal secretion, and severe hypopituitarism
* Patients with impaired liver function
* Patients with untreated hypothyroidism or being treated with drugs that have an action on the hypothalamic-pituitary-adrenal axis
* Patients with hypersensitivity to the active ingredient or any of the excipients listed in section 6.1 of the RCP - Metirapone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-02-17 (Estimated)

PRIMARY OUTCOMES:
Change in Number and/or Dosage of Antihypertensive Drugs at 12 Months with Metirapone Treatment, Maintaining Target Blood Pressure Range | through study completion, an average of 2 months
  This measure will assess any change in the number or dosage of antihypertensive medications required after 12 months of treatment with Metirapone, while maintaining the target blood pressure range (BP >100/60 mmHg and <130/85 mmHg).

SECONDARY OUTCOMES:
"Concentration of Key Biomarkers in Plasma for Monitoring Efficacy of Metirapone Therapy | through study completion, an average of 2 months
  This outcome measure evaluates the efficacy of Metirapone therapy by quantifying the concentration of specific biomarkers in plasma.
  Each biomarker will be measured at predefined time points during the study to monitor changes over time and assess therapeutic response. The values for each biomarker will be reported separately to ensure clarity in units of measure and clinical significance.
"Assessment of Changes in Adrenal Gland Morphology Following Metirapone Therapy | through study completion, an average of 2 months
  This outcome measure evaluates morphological changes in the adrenal glands after treatment with Metirapone. Changes will be summarized as mean differences in adrenal gland size and percentage of participants showing notable structural changes.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Di Dalmazi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (3):
- Italy (3):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedale-Università Padova, Padua